CLINICAL TRIAL: NCT04613999
Title: A Phase 1 Open-label, Non-randomized, Single Ascending Dose Escalation Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of A Ralinepag Extended Release (XR) Tablet Formulation In Healthy Chinese Subjects
Brief Title: A Study of Ralinepag in Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Everstar Medicines (Shanghai) Limited (Industry)
Responsible Party: Sponsor
Organization: Everstar Therapeutics Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES102102
Record Dates: First submitted 2020-09-30; First posted 2020-11-03 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteer; Pharmacokinetic Study
Keywords: Healthy volunteer; Pharmacokinetic, safety and tolerability; Ralinepag
MeSH Terms: interventions — ralinepag

STUDY DESIGN:
Intervention Model Description: The study is planned to enroll 15 subjects with open-label, fixed sequence, non-randomized to take a single dose of ralinepag at 3 separate dose intervals. Ralinepag will be administered at doses of 50, 100 and 150 mcg single oral each time. Subjects will receive Regimen A (single dose of ralinepag 50 mcg) in the morning of Day 1 and pharmacokinetic assessments will be conducted pre-dose and over the 96 hours post-dose. There will be a washout period of 7 days between each IMP administration. Regimens B and C (single dose of ralinepag 100 mcg and ralinepag 150 mcg) will be administered following an overnight fast on Day 8 and 15, respectively, with 96 hours of pharmacokinetic assessments as performed with Regimen A. A Follow-up phone call will take place 10±1 days post-last dose to ensure the ongoing well-being of the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Subjects will receive regimens 50 mcg, 100 mcg and 150 mcg in a sequential manner in consecutive treatment periods. Subjects who have tolerated the IMP in all prior regimens will continue in the study to receive each subsequent dose.
  Interventions: Drug: Ralinepag

INTERVENTIONS:
Drug: Ralinepag — Ralinepag will be supplied as 50 mcg round, orange, XR tablets for oral administration.
  It is planned that every subject will receive each of the following regimens in the fasted state:
  * Regimen A (50 mcg): 1 × 50 mcg ralinepag XR tablet
  * Regimen B (100 mcg): 2 × 50 mcg ralinepag XR tablets
  * Regimen C (150 mcg): 3 × 50 mcg ralinepag XR tablets Subjects will receive Regimens A, B and C in a sequential manner in consecutive treatment periods. Subjects who have tolerated the IMP in all prior regimens will continue in the study to receive each subsequent dose.

SUMMARY:
A Phase 1 Open-label, Non-randomized, Single Ascending Dose Escalation Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of A Ralinepag Extended Release (XR) Tablet Formulation In Healthy Chinese Subjects.

DETAILED DESCRIPTION:
This is a single center, open-label, fixed sequence, non-randomized study of healthy subjects. The study is planned to enroll 15 subjects to ensure data for 8 evaluable subjects.

Subjects will visit the clinical unit for a screening visit up to 28 days before dosing. Eligible subjects will be admitted to the clinical unit prior to investigational medicinal product (IMP) administration (Day -1) and will remain onsite through the study discharge on Day 19. Following an overnight fast of at least 8 hours, subjects will receive Regimen A (single dose of ralinepag 50 mcg) in the morning of Day 1 and pharmacokinetic assessments will be conducted pre-dose and over the 96 hours post-dose. There will be a washout period of 7 days between each IMP administration. Regimens B and C (single dose of ralinepag 100 mcg and ralinepag 150 mcg) will be administered following an overnight fast on Day 8 and 15, respectively, with 96 hours of pharmacokinetic assessments as performed with Regimen A. A Follow-up phone call will take place 10±1 days post-last dose to ensure the ongoing well-being of the subjects. Ralinepag (APD811) will be supplied as 50 mcg round, orange, XR tablets for oral administration.

It is planned that every subject will receive each of the following regimens in the fasted state:

* Regimen A (50 mcg): 1 × 50 mcg ralinepag XR tablet
* Regimen B (100 mcg): 2 × 50 mcg ralinepag XR tablets
* Regimen C (150 mcg): 3 × 50 mcg ralinepag XR tablets Subjects will receive Regimens A, B and C in a sequential manner in consecutive treatment periods. Subjects who have tolerated the IMP in all prior regimens will continue in the study to receive each subsequent dose.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy subjects aged 18 to 45 years at the time of signing the informed consent form (ICF).

  2. Body mass index of 19.0 to 25.0 kg/m2.

  3. In good general health, free from clinically significant medical or psychiatric illness or disease (as determined by medical/surgical history, physical examination, weight, 12-lead ECG and clinical laboratory tests).

  4. HIV, Syphilitics, Hepatitis B and Hepatitis C negative at the screening evaluation.

  5. Adequate venous access in the left or right arm to allow for collection of a number of blood samples

  6. Provides written informed consent.

  7. Willing to comply with all study procedures and requirements.

  8. Subjects of reproductive potential must agree to use an approved method of contraception from Day -1 until 30 days after study discharge:
  1. Barrier method (e.g., condom) plus an approved method of highly effective contraception or
  2. Female/male partner is surgically sterile.

     Exclusion Criteria:
* 1. History or presence of malignancy, with the exception of adequately treated localized skin cancer (basal cell or squamous cell carcinoma), which is allowed.

  2. History or presence of any clinically significant psychiatric condition (including depression or prior suicidal behaviour).

  3. Evidence of clinically relevant medical illness, cardiovascular, hematological, gastrointestinal, hepatic, renal, rheumatologic, endocrine, pulmonary, neurologic, psychiatric or skin disorder (excluding skin cancer as described in Exclusion Criterion 1) or history of hypertension or heart disease including any abnormal laboratory results deemed clinically significant by the study investigator at screening.

  4. History of dysphagia.

  5. Clinically significant surgical procedure or traumatic injury within 3 months of screening.

  6. History of epilepsy (other than febrile seizures during childhood).

  7. Clinically significant infection within 28 days of start of dosing.

  8. Currently suffers from clinically significant systemic allergic disease or has a history of significant drug allergies including a history of anaphylactic reaction (particularly reactions to general anesthetic agents); allergic reaction due to any drug which led to significant morbidity.

  9. History or presence of cardiac arrhythmia or congenital long QT syndrome.

  10. QTcF >450 msec, PR >220 msec and QRS >120 msec on screening ECG (ECG may be repeated after consultation with the Medical Monitor).

  11. Use of tobacco or nicotine containing products in the previous 6 months prior to dosing or use of a nicotine patch within 14 days prior to screening.

  12. Regular alcohol consumption > 2 units/day (1 unit = 300 mL of beer or 45 mL of alcohol 40% or 150mL of wine) or alcohol consumption within 48 hours of start of dosing.

  13. Positive urine drug or alcohol breathalyzer test prior to study entry or history of alcohol or drug abuse in the last 12 months.

  14. Use of any prescription medication within 14 days prior to screening.

  15. Use of any over the counter (OTC) medication, herbal or hormone supplements, or diet aids within 14 days prior to screening

  16. Participation in any other investigational trial in which the last dose of study drug occurred within 30 days or 5 half-lives (whichever is longer) before Check-in for Inpatient Period (Day -1)

  17. Donation of blood from 30 days before Check-in for Inpatient Period (Day -1) or of plasma from 2 weeks before Check-in for Inpatient Period (Day -1)

  18. Receipt of blood products within 2 months before Check-in for Inpatient Period (Day -1)

  19. Abnormal supine BP (defined as either systolic BP > 140 millimetres (mm) Hg or < 90 mmHg or diastolic BP > 90 mmHg or < 50 mmHg) or abnormal pulse rate (> 100 beats per minute [bpm] or < 50 bpm), confirmed by at least 1 repeat measurement

  20. Abnormal orthostatic BP at Screening or CPC Check-in on Day -1 (defined as confirmed drop in SBP > 20 mmHg or drop in DBP > 10 mmHg with standing). The assessment may be repeated once to assure adequate hydration.

  21. Women who are pregnant, lactating or breast-feeding.

  22. Known hypersensitivity to any of the excipients of Ralinepag.

  23. Any inappropriate condition to participate in the study considered by investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Cmax | Baseline to 96 hours
  Maximum concentration determined directly from the concentration-time profile
Tmax | Baseline to 96 hours
  Time to maximum concentration determined directly from the concentration-time profile
T1/2 | Baseline to 96 hours
  Terminal elimination half-life calculated as: ln2/λz
AUC0-24 | Baseline to 96 hours
  Area under the concentration-time curve (AUC) from pre-dose (time 0) to 24 hours post-dose calculated using the linear-log trapezoidal rule
AUClast | Baseline to 96 hours
  AUC from time zero to the time of the last quantifiable concentration (Tlast) calculated using the linear-log trapezoidal rule
AUCinf | Baseline to 96 hours
  AUC from pre-dose (Time 0) extrapolated to infinite time (AUClast + Clast/λz) calculated using the linear-log trapezoidal rule

SECONDARY OUTCOMES:
Adverse event reporting | From signing ICF to 10 days after last dose.
Assessment of general appearance of dermatologic. | From signing ICF to 10 days after last dose.
Assessment of general appearance of head. | From signing ICF to 10 days after last dose.
Assessment of general appearance of eyes. | From signing ICF to 10 days after last dose.
Assessment of general appearance of ears. | From signing ICF to 10 days after last dose.
Assessment of general appearance of mouth. | From signing ICF to 10 days after last dose.
Assessment of general appearance of throat. | From signing ICF to 10 days after last dose.
Assessment of general appearance of neck. | From signing ICF to 10 days after last dose.
Assessment of general appearance of thyroid. | From signing ICF to 10 days after last dose.
Assessment of general appearance of lymph nodes. | From signing ICF to 10 days after last dose.
Assessment of general appearance of respiratory system. | From signing ICF to 10 days after last dose.
Assessment of general appearance of cardiovascular system. | From signing ICF to 10 days after last dose.
Assessment of general appearance of gastrointestinal system. | From signing ICF to 10 days after last dose.
Assessment of general appearance of extremities. | From signing ICF to 10 days after last dose.
Assessment of general appearance of musculoskeletal system. | From signing ICF to 10 days after last dose.
Assessment of general appearance of neurologic system. | From signing ICF to 10 days after last dose.
Assessment of general appearance of psychiatric system. | From signing ICF to 10 days after last dose.
Serum alanine aminotransferase (ALT) | From signing ICF to 10 days after last dose.
Serum glucose | From signing ICF to 10 days after last dose.
Serum albumin | From signing ICF to 10 days after last dose.
Serum lactate dehydrogenase (LDH) | From signing ICF to 10 days after last dose.
Serum alkaline phosphatase (ALP) | From signing ICF to 10 days after last dose.
Serum phosphorus | From signing ICF to 10 days after last dose.
Serum aspartate aminotransferase (AST) | From signing ICF to 10 days after last dose.
Serum potassium | From signing ICF to 10 days after last dose.
Serum blood urea | From signing ICF to 10 days after last dose.
Serum sodium | From signing ICF to 10 days after last dose.
Serum calcium | From signing ICF to 10 days after last dose.
Serum total bilirubin | From signing ICF to 10 days after last dose.
Serum cholesterol | From signing ICF to 10 days after last dose.
Serum triglycerides | From signing ICF to 10 days after last dose.
Serum creatinine | From signing ICF to 10 days after last dose.
Serum uric acid | From signing ICF to 10 days after last dose.
Serum creatine phosphokinase (CPK) | From signing ICF to 10 days after last dose.
Serum gamma glutamyl transferase (GGT | From signing ICF to 10 days after last dose.
White blood cell (WBC) count | From signing ICF to 10 days after last dose.
Neutrophils (percentage and absolute count) | From signing ICF to 10 days after last dose.
Red blood cell (RBC) count | From signing ICF to 10 days after last dose.
Lymphocytes (percentage） | From signing ICF to 10 days after last dose.
Lymphocytes (absolute count) | From signing ICF to 10 days after last dose.
Hemoglobin (Hb) | From signing ICF to 10 days after last dose.
Monocytes (percentage) | From signing ICF to 10 days after last dose.
Monocytes (absolute count) | From signing ICF to 10 days after last dose.
Hematocrit (HCT) | From signing ICF to 10 days after last dose.
Eosinophils (percentage) | From signing ICF to 10 days after last dose.
Eosinophils (absolute count) | From signing ICF to 10 days after last dose.
Mean corpuscular volume (MCV) | From signing ICF to 10 days after last dose.
Basophils (percentage) | From signing ICF to 10 days after last dose.
Basophils (absolute count) | From signing ICF to 10 days after last dose.
Mean corpuscular hemoglobin (MCH) | From signing ICF to 10 days after last dose.
Platelet count | From signing ICF to 10 days after last dose.
Mean corpuscular hemoglobin concentration (MCHC) | From signing ICF to 10 days after last dose.
RBC distribution width | From signing ICF to 10 days after last dose.
Urine bilirubin | From signing ICF to 10 days after last dose.
Urine blood | From signing ICF to 10 days after last dose.
Urine glucose | From signing ICF to 10 days after last dose.
Urine PH | From signing ICF to 10 days after last dose.
Urine specific gravity | From signing ICF to 10 days after last dose.
Urine ketones | From signing ICF to 10 days after last dose.
Urine protein | From signing ICF to 10 days after last dose.
Urine leukocytes | From signing ICF to 10 days after last dose.
Urine urobilinogen | From signing ICF to 10 days after last dose.
Urine nitrite | From signing ICF to 10 days after last dose.
Urine microscopic (only for abnormal urine stick test findings). | From signing ICF to 10 days after last dose.
Supine BP | From signing ICF to 10 days after last dose.
Pulse | From signing ICF to 10 days after last dose.
Body temperature | From signing ICF to 10 days after last dose.
Respiratory rate | From signing ICF to 10 days after last dose.
ECG PR interval | From signing ICF to 10 days after last dose.
ECG QRS interval | From signing ICF to 10 days after last dose.
ECG RR interval | From signing ICF to 10 days after last dose.
ECG QT interval | From signing ICF to 10 days after last dose.
ECG QT interval corrected for heart rate (QTc) | From signing ICF to 10 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Li, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No